CLINICAL TRIAL: NCT02666664
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Long-term Safety and Tolerability Study of ETC-1002 in Patients With Hyperlipidemia at High Cardiovascular Risk Who Are Not Adequately Controlled by Their Lipid-Modifying Therapy
Brief Title: Evaluation of Long-Term Safety and Tolerability of ETC-1002 in High-Risk Patients With Hyperlipidemia and High CV Risk (CLEAR Harmony)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1002-040; 2015-004136-36 (EudraCT Number)
Record Dates: First submitted 2016-01-20; First posted 2016-01-28 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: Hypercholesterolemia; Atherosclerotic Cardiovascular Diseases
Keywords: hyperlipidemia; cholesterol; heterozygous familial hypercholesterolemia; atherosclerotic cardiovascular disease; ASCVD; HeFH; LDL
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Atherosclerosis | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETC-1002 (Experimental): ETC-1002 180 mg/day
  Interventions: Drug: ETC-1002
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ETC-1002 — ETC-1002 180 mg tablets taken orally, once per day. Patients remain on ongoing statin therapy (not study provided)
  Other Names: bempedoic acid
  Arms: ETC-1002
Drug: Placebo — Matching placebo tablets taken orally, once per day. Patients remain on ongoing statin therapy (not study provided)
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if ETC-1002 (bempedoic acid) is safe and well-tolerated versus placebo in patients with high cardiovascular risk and elevated LDL cholesterol that is not adequately controlled by their current therapy.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-C ≥ 70 mg/dL
* High cardiovascular risk (diagnosis of HeFH or ASCVD)
* Be on maximally tolerated lipid-modifying therapy

Exclusion Criteria:

* Total fasting triglyceride ≥500 mg/dL
* Renal dysfunction or nephrotic syndrome or history of nephritis
* Body Mass Index (BMI) ≥50kg/m2
* Significant cardiovascular disease or cardiovascular event in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2230 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Haberman, MD, Study Director — Esperion Therapeutics, Inc.
Locations (104):
- United States (48):
  - Huntsville, Alabama
  - Cottonwood, Arizona
  - Phoenix, Arizona
  - Canoga Park, California
  - Santa Rosa, California
  - Bridgeport, Connecticut
  - Hartford, Connecticut
  - Atlantis, Florida
  - Boca Raton, Florida
  - Crestview, Florida
  - Crystal River, Florida
  - Daytona Beach, Florida
  - Lake Worth, Florida
  - Miami Lakes, Florida
  - Tampa, Florida
  - Park Ridge, Illinois
  - Iowa City, Iowa
  - Overland Park, Kansas
  - Covington, Kentucky
  - Louisville, Kentucky
  - Minden, Louisiana
  - Monroe, Louisiana
  - Shreveport, Louisiana
  - Auburn, Maine
  - Midland, Michigan
  - Saginaw, Michigan
  - Saint Cloud, Minnesota
  - Tupelo, Mississippi
  - Jefferson City, Missouri
  - Nashua, New Hampshire
  - Bridgewater, New Jersey
  - Cary, North Carolina
  - Mount Airy, North Carolina
  - Raleigh, North Carolina
  - Rocky Mount, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Sandusky, Ohio
  - Willoughby, Ohio
  - Hillsboro, Oregon
  - Fort Worth, Texas
  - Houston, Texas
  - Katy, Texas
  - Kingwood, Texas
  - Orem, Utah
  - Richmond, Virginia
  - Puyallup, Washington
  - Tacoma, Washington
- Canada (14):
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Gatineau, Ontario
  - Mississauga, Ontario
  - Oshawa, Ontario
  - Peterborough, Ontario
  - Scarborough Village, Ontario
  - Chicoutimi, Quebec
  - Gatineau, Quebec
  - Longueuil, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Charles-Borromée, Quebec
  - Saint-Jean-sur-Richelieu, Quebec
- Germany (7):
  - Berlin
  - Bochum
  - Dresden
  - Essen
  - Frankfurt
  - Leipzig
  - München
- Netherlands (11):
  - Amsterdam
  - Arnhem
  - Eindhoven
  - Goes
  - Groningen
  - Hardenberg
  - Leiden
  - Rotterdam
  - Tilburg
  - Venlo
  - Zutphen
- Poland (10):
  - Gdansk
  - Gdynia
  - Katowice
  - Krakow
  - Lodz
  - Lowicz
  - Poznan
  - Puławy
  - Torun
  - Wroclaw
- United Kingdom (14):
  - Bexhill-on-Sea
  - Birmingham
  - Cardiff
  - Chesterfield
  - Chichester
  - Chippenham
  - Chorley
  - Glasgow
  - Hexham
  - Hull
  - Ipswich
  - Liverpool
  - Manchester
  - Reading

REFERENCES:
- [Background] Pinkosky SL, Newton RS, Day EA, Ford RJ, Lhotak S, Austin RC, Birch CM, Smith BK, Filippov S, Groot PHE, Steinberg GR, Lalwani ND. Liver-specific ATP-citrate lyase inhibition by bempedoic acid decreases LDL-C and attenuates atherosclerosis. Nat Commun. 2016 Nov 28;7:13457. doi: 10.1038/ncomms13457. PMID 27892461
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Background] Goldberg AC, Hopkins PN, Toth PP, Ballantyne CM, Rader DJ, Robinson JG, Daniels SR, Gidding SS, de Ferranti SD, Ito MK, McGowan MP, Moriarty PM, Cromwell WC, Ross JL, Ziajka PE; National Lipid Association Expert Panel on Familial Hypercholesterolemia. Familial hypercholesterolemia: screening, diagnosis and management of pediatric and adult patients: clinical guidance from the National Lipid Association Expert Panel on Familial Hypercholesterolemia. J Clin Lipidol. 2011 Jun;5(3 Suppl):S1-8. doi: 10.1016/j.jacl.2011.04.003. Epub 2011 Apr 12. PMID 21600525
- [Background] Pollex RL, Joy TR, Hegele RA. Emerging antidyslipidemic drugs. Expert Opin Emerg Drugs. 2008 Jun;13(2):363-81. doi: 10.1517/14728214.13.2.363. PMID 18537526
- [Background] Sharrett AR, Ballantyne CM, Coady SA, Heiss G, Sorlie PD, Catellier D, Patsch W; Atherosclerosis Risk in Communities Study Group. Coronary heart disease prediction from lipoprotein cholesterol levels, triglycerides, lipoprotein(a), apolipoproteins A-I and B, and HDL density subfractions: The Atherosclerosis Risk in Communities (ARIC) Study. Circulation. 2001 Sep 4;104(10):1108-13. doi: 10.1161/hc3501.095214. PMID 11535564
- [Result] Ray KK, Bays HE, Catapano AL, Lalwani ND, Bloedon LT, Sterling LR, Robinson PL, Ballantyne CM; CLEAR Harmony Trial. Safety and Efficacy of Bempedoic Acid to Reduce LDL Cholesterol. N Engl J Med. 2019 Mar 14;380(11):1022-1032. doi: 10.1056/NEJMoa1803917. PMID 30865796
- [Derived] Ridker PM, Lei L, Ray KK, Ballantyne CM, Bradwin G, Rifai N. Effects of bempedoic acid on CRP, IL-6, fibrinogen and lipoprotein(a) in patients with residual inflammatory risk: A secondary analysis of the CLEAR harmony trial. J Clin Lipidol. 2023 Mar-Apr;17(2):297-302. doi: 10.1016/j.jacl.2023.02.002. Epub 2023 Feb 14. PMID 36813656
- [Derived] Ballantyne CM, Bays HE, Louie MJ, Smart J, Zhang Y, Ray KK. Factors Associated With Enhanced Low-Density Lipoprotein Cholesterol Lowering With Bempedoic Acid. J Am Heart Assoc. 2022 Aug 2;11(15):e024531. doi: 10.1161/JAHA.121.024531. Epub 2022 Aug 2. PMID 35916348
- [Derived] Banach M, Duell PB, Gotto AM Jr, Laufs U, Leiter LA, Mancini GBJ, Ray KK, Flaim J, Ye Z, Catapano AL. Association of Bempedoic Acid Administration With Atherogenic Lipid Levels in Phase 3 Randomized Clinical Trials of Patients With Hypercholesterolemia. JAMA Cardiol. 2020 Oct 1;5(10):1124-1135. doi: 10.1001/jamacardio.2020.2314. PMID 32609313
- See also: World Health Organization Fact Sheet No. 317 — http://www.who.int/mediacentre/factsheets/fs317/en/
- See also: Familial Hypercholesterolemia Foundation — https://thefhfoundation.org/familial-hypercholesterolemia/what-is-familial-hypercholesterolemia
- See also: National Organization for Rare Disorders - Familial Hypercholesterolemia — https://rarediseases.org/rare-diseases/familial-hypercholesterolemia/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2230 participants were randomized 2:1 to either bempedoic acid or placebo. One participant was randomized to bempedoic acid treatment, but never received any dose of investigational medicinal product (IMP) i.e. study drug.
Pre-assignment Details: The study consisted of 2 periods: a 2-week screening period and a 52-week double-blind, randomized treatment period.
Groups:
- Placebo: During the double-blind treatment period, participants received placebo tablet, once daily by mouth for 52 weeks. In addition, participants received stable background lipid-modifying therapy(ies) including a maximally tolerated statin throughout the study.
- Bempedoic Acid: During the double-blind treatment period, participants received bempedoic acid 180 mg tablet, once daily by mouth for 52 weeks. In addition, participants received stable background lipid-modifying therapy(ies) including a maximally tolerated statin throughout the study.
Period: Overall Study
Arm/Group | Placebo | Bempedoic Acid
Started | 742 | 1488
Completed | 706 | 1404
Not Completed | 36 | 84
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Other | 0 | 1
Not completed — Adverse Event | 12 | 37
Not completed — Withdrawal by participant | 23 | 40
Not completed — Sponsor decision | 0 | 1
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bempedoic Acid | Total
Number analyzed (Participants) | 742 | 1488 | 2230
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (8.64) | 65.8 (9.11) | 66.1 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 389 | 602
  Male | 529 | 1099 | 1628
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 24 | 35
  Not Hispanic or Latino | 731 | 1464 | 2195
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 8 | 14 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 15 | 42 | 57
  White | 716 | 1423 | 2139
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 4 | 6
Cardiovascular history: atherosclerotic cardiovascular disease (ASCVD) [Count of Participants; unit: Participants]
  Yes | 727 | 1449 | 2176
  No | 15 | 39 | 54
Cardiovascular history: heterozygous familial hypercholesterolemia (HeFH) [Count of Participants; unit: Participants]
  Yes | 23 | 56 | 79
  No | 719 | 1432 | 2151
History of diabetes [Count of Participants; unit: Participants]
  Yes | 212 | 425 | 637
  No | 530 | 1063 | 1593
History of hypertension [Count of Participants; unit: Participants]
  Yes | 594 | 1174 | 1768
  No | 148 | 314 | 462
Concomitant lipid-modifying therapy (LMT): Statin [Count of Participants; unit: Participants] — Concomitant medications are defined as medications that were ongoing at the time of double-blind study drug initiation or new medications that started post double-blind study drug initiation and within 30 days following the date of the last dose of study drug.
  Participants
    Yes | 742 | 1485 | 2227
    No | 0 | 3 | 3
Concomitant LMT: Ezetimibe [Count of Participants; unit: Participants] — Concomitant medications are defined as medications that were ongoing at the time of double-blind study drug initiation or new medications that started post double-blind study drug initiation and within 30 days following the date of the last dose of study drug.
  Participants
    Yes | 56 | 116 | 172
    No | 686 | 1372 | 2058
Concomitant LMT: Fibrate [Count of Participants; unit: Participants] — Concomitant medications are defined as medications that were ongoing at the time of double-blind study drug initiation or new medications that started post double-blind study drug initiation and within 30 days following the date of the last dose of study drug.
  Participants
    Yes | 26 | 54 | 80
    No | 716 | 1434 | 2150
Concomitant LMT: None [Count of Participants; unit: Participants] — Concomitant medications are defined as medications that were ongoing at the time of double-blind study drug initiation or new medications that started post double-blind study drug initiation and within 30 days following the date of the last dose of study drug.
  Participants
    Concomitant LMT: None | 0 | 2 | 2
    Concomitant LMT: Yes | 742 | 1486 | 2228
Baseline statin intensity [Count of Participants; unit: Participants] — Baseline statin intensity were based on stratification at randomization. Low-intensity statins: simvastatin 10 milligrams (mg); pravastatin 10-20 mg; lovastatin 20 mg; fluvastatin 20-40 mg; pitavastatin 1 mg. Moderate-intensity statins: atorvastatin 10-20 mg; rosuvastatin 5-10 mg; simvastatin 20 mg; pravastatin 40-80 mg; lovastatin 40 mg; fluvastatin XL 80 mg; fluvastatin 40 mg twice a day; pitavastatin 2-4 mg. High-intensity statins: atorvastatin 40-80 mg; rosuvastatin 20-40 mg.
  Participants
    Low | 48 | 100 | 148
    Moderate | 324 | 646 | 970
    High | 370 | 742 | 1112
Estimated glomerular filtration rate (eGFR) [Count of Participants; unit: Participants] — milliliter per minute per 1.73 square meter = ml/min/1.73m^2
  Participants
    Normal: ≥ 90 mL/min/1.73m^2 | 167 | 320 | 487
    Mild Renal Impairment: 60-89 mL/min/1.73m^2 | 468 | 946 | 1414
    Moderate Renal Impairment: 30-59 mL/min/1.73m^2 | 107 | 222 | 329
Total cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1).
  mg/dL | 178.64 (35.645) | 179.66 (35.143) | 179.32 (35.306)
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1).
  mg/dL | 102.30 (30.048) | 103.60 (29.127) | 103.16 (29.436)
High-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1).
  mg/dL | 49.29 (11.545) | 48.71 (11.853) | 48.90 (11.752)
Triglycerides (TG) [Median (Inter-Quartile Range); unit: mg/dL] — Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1).
  mg/dL | 122.50 [95.50 to 169.50] | 126.25 [98.00 to 165.50] | 125.00 [97.50 to 167.00]
Non-high-density lipoprotein cholesterol (non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1).
  mg/dL | 129.37 (33.855) | 130.92 (33.677) | 130.41 (33.737)
Apolipoprotein B (apoB) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the last value prior to first dose of study drug.
  mg/dL | 86.8 (21.82) | 88.5 (21.57) | 87.9 (21.66)
High-sensitivity C-reactive protein (hsCRP) [Median (Inter-Quartile Range); unit: mg/L] — Baseline was defined as the last value prior to the first dose of study drug.
  mg/L | 1.51 [0.79 to 3.33] | 1.49 [0.74 to 3.28] | 1.49 [0.76 to 3.30]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs, defined as adverse events (AEs) that began or worsened in severity after the first dose of double-blind study drug and up to 30 days after receiving the last dose of double-blind study drug, were collected and reported.
Time Frame: Up to approximately 52 weeks
Population: Safety Population: all randomized participants who received at least 1 dose of investigational medicinal product. Participants were included in the treatment group that they received, regardless of their randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
percentage of participants
  Any TEAE | 78.7 | 78.5
  Any serious TEAE | 14.0 | 14.5
  Any fatal TEAE | 0.3 | 0.9
  Any TEAE leading to discontinuation of study drug | 7.1 | 10.9

2. Primary Outcome: Percentage of Participants With Adjudicated Major Adverse Cardiovascular Event
Description: TEAEs, defined as AEs that began or worsened in severity after the first dose of double-blind study drug and up to 30 days after receiving the last dose of double-blind study drug, were collected and reported. Cardiovascular events were considered as adverse events of special interest. Treatment-emergent = TE.
Time Frame: Up to approximately 52 weeks
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
percentage of participants
  Any adjudicated major clinical event | 5.7 | 4.6
  Any TE death from cardiovascular causes | 0.1 | 0.4
  Any nonfatal myocardial infarction | 1.8 | 1.3
  Any nonfatal stroke | 0.3 | 0.3
  Any coronary revascularization | 3.2 | 2.6
  Any hospitalization for unstable angina | 1.5 | 0.9
  TE death from noncardiovascular causes | 0.1 | 0.1
  Noncoronary arterial revascularization | 0.8 | 0.3
  Hospitalization for heart failure | 0.1 | 0.6

3. Primary Outcome: Percentage of Participants With the Indicated Event of Special Interest: Creatine Kinase Elevations
Description: TEAEs of special interest (AESIs) were predefined and monitored throughout the study. Creatine kinase elevations were assessed using the following preferred term: Blood creatine phosphokinase increased (system organ class: investigations).
Time Frame: Up to approximately 52 weeks
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
percentage of participants | 1.8 | 2.4

4. Primary Outcome: Percentage of Participants With the Indicated Event of Special Interest: Hepatic Disorders
Description: Treatment-emergent AESIs were predefined and monitored throughout the study. TEAEs potentially related to hepatic events were assessed using the following preferred terms and laboratory abnormalities: aspartate aminotransferase (AST) increased, Alanine aminotransferase (ALT) increased, Hepatic enzyme increased, Blood bilirubin increased, liver function test (LFT) abnormal, LFT increased, hepatic enzyme abnormal, transaminases increased, potential Hy's Law cases (PHLC) [AST and (&)/or ALT >3 x upper limit of normal (ULN) with concurrent total bilirubin >2 x ULN], AST and/or ALT >3 x ULN, and total bilirubin >2 x ULN (system organ class: investigations). AST and ALT values were repeated and confirmed. "Repeated and confirmed" was defined as a participant having the last on-study LFT > x ULN, the last on-treatment LFT > x ULN, or LFT > x ULN followed by another LFT > x ULN.
Time Frame: Up to approximately 52 weeks
Population: Safety Population. The percentage of unique participants is reported in the "Overall hepatic disorder AESIs" category; a participant could have been represented in more than one of the individual hepatic disorder AESIs.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
percentage of participants
  Overall hepatic disorder AESIs | 1.5 | 2.5
  AST increased | 0.4 | 1.5
  ALT increased | 0.3 | 0.8
  Hepatic enzyme increased | 0.0 | 0.5
  Blood bilirubin increased | 0.4 | 0.1
  Liver function test abnormal | 0.3 | 0.1
  Liver function test increased | 0.1 | 0.2
  Hepatic enzyme abnormal | 0.0 | 0.1
  Transaminases increased | 0.1 | 0.0
  PHLC [AST &/or ALT>3 x ULN, concurrent TB>2 x ULN] | 0.0 | 0.0
  AST and/or ALT >3 x ULN | 0.1 | 0.5
  Total bilirubin >2 x ULN | 0.0 | 0.0

5. Primary Outcome: Percentage of Participants With the Indicated Event of Special Interest: Hypoglycemia
Description: Treatment-emergent AESIs were predefined and monitored throughout the study. Hypoglycemia was assessed using the following preferred terms: hypoglycaemia (system organ class: metabolism and nutrition disorders); blood glucose abnormal and blood glucose decreased (system organ class: investigations). The percentage of unique participants is reported in the "Overall hypoglycemia AESIs" category; a participant could have been represented in more than one of the individual hypoglycemia AESIs.
Time Frame: Up to approximately 52 weeks
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
percentage of participants
  Overall hypoglycemia AESIs | 3.1 | 2.2
  Hypoglycaemia | 3.0 | 2.2
  Blood glucose abnormal | 0.1 | 0.1
  Blood glucose decreased | 0.0 | 0.1

6. Primary Outcome: Percentage of Participants With the Indicated Event of Special Interest: Metabolic Acidosis
Description: Treatment-emergent AESIs were predefined and monitored throughout the study. Metabolic acidosis was assessed using the preferred term metabolic acidosis (system organ class: metabolism and nutrition disorders).
Time Frame: Up to approximately 52 weeks
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
percentage of participants | 0.0 | 0.1

7. Primary Outcome: Percentage of Participants With the Indicated Event of Special Interest: Muscular Disorder
Description: Treatment-emergent AESIs were predefined and monitored throughout the study. Muscular safety was assessed using the following preferred terms and laboratory abnormalities: myalgia, muscle spasms, pain in extremity, muscular weakness (system organ class: musculoskeletal and connective tissue disorders), and creatine kinase >5 ULN (repeated and confirmed). The percentage of unique participants is reported in the "Overall muscular disorder AESIs" category; a participant could have been represented in more than one of the individual muscular disorder AESIs.
Time Frame: Up to approximately 52 weeks
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
percentage of participants
  Overall muscular disorder AESIs | 10.1 | 13.1
  Myalgia | 6.1 | 6.0
  Muscle spasms | 2.7 | 4.2
  Pain in extremity | 2.2 | 3.4
  Muscular weakness | 0.5 | 0.6
  Creatine kinase >5 ULN | 0.1 | 0.5

8. Primary Outcome: Percentage of Participants With the Indicated Event of Special Interest: Neurocognitive Disorder
Description: Treatment-emergent AESIs were predefined and monitored throughout the study. Neurocognitive disorder was assessed using the following preferred terms: memory impairment, amnesia, and cognitive disorder (system organ class: nervous system disorders); confusional state and disorientation (system organ class: psychiatric disorders). The percentage of unique participants is reported in the "Overall neurocognitive disorder AESIs" category; a participant could have been represented in more than one of the individual neurocognitive disorder AESIs.
Time Frame: Up to approximately 52 weeks
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
percentage of participants
  Overall neurocognitive disorder AESIs | 0.9 | 0.7
  Memory impairment | 0.5 | 0.3
  Amnesia | 0.4 | 0.2
  Cognitive disorder | 0.0 | 0.1
  Confusional state | 0.0 | 0.1
  Disorientation | 0.0 | 0.1

9. Primary Outcome: Percentage of Participants With the Indicated Event of Special Interest: New Onset or Worsening Diabetes Mellitus
Description: Treatment-emergent AESIs were predefined and monitored throughout the study. New onset or worsening diabetes was assessed using the following preferred terms: type 2 diabetes mellitus, diabetes mellitus, hyperglycaemia, glucose tolerance impaired, diabetes mellitus inadequate control, and impaired fasting glucose (system organ class: metabolism and nutrition disorders); blood glucose increased, glycosylated haemoglobin increased, blood glucose abnormal, and glucose urine present (system organ class: investigations); and glycosuria (system organ class: renal and urinary disorders). The percentage of unique participants is reported in the "Overall new onset/worsening diabetes mellitus AESIs" category; a participant could have been represented in more than one of the individual new onset/worsening diabetes mellitus AESIs.
Time Frame: Up to approximately 52 weeks
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
percentage of participants
  Overall new onset/worsening diabetes mellitus AESI | 5.4 | 3.3
  Type 2 diabetes mellitus | 0.9 | 1.0
  Diabetes mellitus | 0.9 | 0.4
  Hyperglycaemia | 0.7 | 0.5
  Glucose tolerance impaired | 0.1 | 0.4
  Diabetes mellitus inadequate control | 0.4 | 0.1
  Impaired fasting glucose | 0.3 | 0.1
  Blood glucose increased | 1.2 | 0.7
  Glycosylated haemoglobin increased | 0.5 | 0.0
  Blood glucose abnormal | 0.1 | 0.1
  Glucose urine present | 0.1 | 0.0
  Glycosuria | 0.3 | 0.1

10. Primary Outcome: Percentage of Participants With the Indicated Event of Special Interest: Renal Disorder
Description: Treatment-emergent AESIs were predefined and monitored throughout the study. TEAEs potentially related to renal events were assessed using the following preferred terms: renal failure, renal impairment, acute kidney injury (system organ class: renal and urinary disorders); blood creatinine increased, glomerular filtration rate decreased, blood urea increased, estimated glomerular filtration rate (eGFR) <30 milliliter per minute per 1.73 square meter (ml/min/1.73m^2), and change from baseline in creatinine >1 mg/dL (system organ class: investigations); and gout (system organ class: metabolism and nutrition disorders). The percentage of unique participants is reported in the "Overall renal disorder AESIs" category; a participant could have been represented in more than one of the individual renal disorder AESIs.
Time Frame: Up to approximately 52 weeks
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
percentage of participants
  Renal failure | 0.1 | 0.9
  Renal impairment | 0.1 | 0.4
  Acute kidney injury | 0.3 | 0.3
  Blood creatinine increased | 0.4 | 0.8
  Glomerular filtration rate decreased | 0.0 | 0.5
  Blood urea increased | 0.1 | 0.1
  Gout | 0.3 | 1.2
  Change from baseline in creatinine >1 mg/dL | 0.0 | 0.1
  eGFR <30 mL/min/1.73 m^2 | 0.4 | 0.9

11. Primary Outcome: Change From Baseline to Week 52 in Uric Acid (Urate) Level
Description: Blood samples were drawn at defined time points during the course of the study to monitor uric acid (urate) levels.
Time Frame: Baseline and Week 52
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
milligrams per deciliter (mg/dL)
  Baseline | 5.96 (1.35) | 6.06 (1.37)
  Change from Baseline at Week 52: number analyzed (Participants) | 680 | 1358
  Change from Baseline at Week 52 | -0.06 (0.87) | 0.73 (1.11)

12. Primary Outcome: Change From Baseline to Week 52 in Creatinine Level
Description: Blood samples were drawn at defined time points during the course of the study to monitor creatinine levels.
Time Frame: Baseline and Week 52
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
mg/dL
  Baseline | 0.96 (0.22) | 0.97 (0.22)
  Change from Baseline at Week 52: number analyzed (Participants) | 677 | 1343
  Change from Baseline at Week 52 | -0.02 (0.12) | 0.02 (0.13)

13. Primary Outcome: Change From Baseline to Week 52 in Hemoglobin Level
Description: Blood samples were drawn at defined time points during the course of the study to monitor hemoglobin levels.
Time Frame: Baseline and Week 52
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1487
grams per deciliter (g/dL)
  Baseline | 14.07 (1.26) | 14.22 (1.26)
  Change from Baseline at Week 52: number analyzed (Participants) | 669 | 1334
  Change from Baseline at Week 52 | -0.23 (0.85) | -0.58 (0.88)

14. Secondary Outcome: Percent Change From Baseline to Week 12 in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for LDL-C. Baseline was defined as the mean of the values at screening (Week -2) and predose Day 1/Week 0. Percent change from baseline was calculated as: [(LDL-C value at Week 12 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Missing data were imputed with the use of a pattern-mixture model to account for adherence to the trial regimen. Least Square mean= LS mean. Percent change was analyzed using the analysis of covariance (ANCOVA) method, which included treatment, randomization stratum as factors, and baseline value as covariate.
Time Frame: Baseline; Week 12
Population: Full Analysis Set: all randomized participants
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1488
percent change | 1.6 (0.86) | -16.5 (0.52)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -18.1, 95% CI 2-sided [-20 to -16.1], Standard Error of Mean 1.01

15. Secondary Outcome: Absolute Change From Baseline to Week 12 in LDL-C
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for LDL-C. Baseline was defined as the mean of the values at screening (Week -2) and predose Day 1/Week 0. Absolute change from baseline was calculated as: LDL-C value at Week 12 minus Baseline value. Missing data were imputed with the use of a pattern-mixture model to account for adherence to the trial regimen.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 725 | 1424
mg/dL | 0.43 (27.04) | -19.23 (24.01)

16. Other Pre Specified Outcome: Percent Change From Baseline to Week 24 in LDL-C
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for LDL-C. Baseline was defined as the mean of the values at screening (Week -2) and predose Day 1/Week 0. Percent change from baseline was calculated as: [(LDL-C value at Week 24 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Missing data were imputed with the use of a pattern-mixture model to account for adherence to the trial regimen. Percent change was analyzed using the ANCOVA method, which included treatment, randomization stratum as factors, and baseline value as covariate.
Time Frame: Baseline; Week 24
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1488
percent change | 1.2 (0.88) | -14.9 (0.60)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -16.1, 95% CI 2-sided [-18.2 to -14], Standard Error of Mean 1.07

17. Other Pre Specified Outcome: Percent Change From Baseline to Week 12 in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for non-HDL-C. Baseline was defined as the mean of the values at screening (Week -2) and predose Day 1/Week 0. Percent change from baseline was calculated as: [(non-HDL-C value at Week 12 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Missing data were imputed with the use of a pattern-mixture model to account for adherence to the trial regimen. Percent change was analyzed using the ANCOVA method, which included treatment, randomization stratum as factors, and baseline value as covariate.
Time Frame: Baseline; Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1488
percent change | 1.5 (0.76) | -11.9 (0.48)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -13.3, 95% CI 2-sided [-15.1 to -11.6], Standard Error of Mean 0.9

18. Other Pre Specified Outcome: Percent Change From Baseline to Week 12 in Total Cholesterol (TC)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for TC. Baseline was defined as the mean of the values at screening (Week -2) and predose Day 1/Week 0. Percent change from baseline was calculated as: [(TC value at Week 12 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Missing data were imputed with the use of a pattern-mixture model to account for adherence to the trial regimen. Percent change was analyzed using the ANCOVA method, which included treatment, randomization stratum as factors, and baseline value as covariate.
Time Frame: Baseline; Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1488
percent change | 0.8 (0.57) | -10.3 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -11.1, 95% CI 2-sided [-12.5 to -9.8], Standard Error of Mean 0.69

19. Other Pre Specified Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein B (apoB)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for apoB. Baseline was defined as the last value prior to first dose of study drug. Percent change from baseline was calculated as: [(apoB value at Week 12 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Missing data were imputed with the use of a pattern-mixture model to account for adherence to the trial regimen. Percent change was analyzed using the ANCOVA method, which included treatment, randomization stratum as factors, and baseline value as covariate.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 736 | 1485
percent change | 3.3 (0.70) | -8.6 (0.47)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -11.9, 95% CI 2-sided [-13.6 to -10.2], Standard Error of Mean 0.85

20. Other Pre Specified Outcome: Percent Change From Baseline to Week 12 in High-sensitivity C-reactive Protein (hsCRP)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for hsCRP. Baseline was defined as the last value prior to first dose of study drug. Percent change from baseline was calculated as: [(hsCRP value at Week 12 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Observed data was used for the analysis, no imputation for the missing data was performed. Percent change was analyzed using the ANCOVA method, which included treatment, randomization stratum as factors, and baseline value as covariate.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 724 | 1421
percent change | 2.6 (91.9) | -22.4 (72.5)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Location shift = -21.5, 95% CI 2-sided [-26.96 to -16], Standard Error of Mean 2.8

21. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in LDL-C
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for LDL-C. Baseline was defined as the mean of the values at screening (Week -2) and predose Day 1/Week 0. Percent change from baseline was calculated as: [(LDL-C value at Week 52 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Observed data was used for the analysis, no imputation for the missing data was performed. Percent change was analyzed using the ANCOVA method, which included treatment, randomization stratum as factors, and baseline value as covariate.
Time Frame: Baseline; Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 685 | 1364
percent change | 1.0 (0.92) | -12.6 (0.66)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -13.6, 95% CI 2-sided [-15.8 to -11.3], Standard Error of Mean 1.13

22. Other Pre Specified Outcome: Percent Change From Baseline to Week 24 in Non-HDL-C
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for non-HDL-C. Baseline was defined as the mean of the values at screening (Week -2) and predose Day 1/Week 0. Percent change from baseline was calculated as: [(non-HDL-C value at Week 24 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Observed data was used for the analysis, no imputation for the missing data was performed.
Time Frame: Baseline; Week 24
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 707 | 1396
percent change | 1.61 (20.91) | -11.69 (19.80)

23. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in Non-HDL-C
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for non-HDL-C. Baseline was defined as the mean of the values at screening (Week -2) and predose Day 1/Week 0. Percent change from baseline was calculated as: [(non-HDL-C value at Week 52 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Observed data was used for the analysis, no imputation for the missing data was performed.
Time Frame: Baseline; Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 685 | 1364
percent change | 0.65 (21.438) | -10.07 (22.097)

24. Other Pre Specified Outcome: Percent Change From Baseline to Week 24 in TC
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for TC. Baseline was defined as the mean of the values at screening (Week -2) and predose Day 1/Week 0. Percent change from baseline was calculated as: [(TC value at Week 24 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Observed data was used for the analysis, no imputation for the missing data was performed.
Time Frame: Baseline; Week 24
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 708 | 1396
percent change | 1.15 (15.349) | -9.86 (15.358)

25. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in TC
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for TC. Baseline was defined as the mean of the values at screening (Week -2) and predose Day 1/Week 0. Percent change from baseline was calculated as: [(TC value at Week 52 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Observed data was used for the analysis, no imputation for the missing data was performed.
Time Frame: Baseline; Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 685 | 1365
percent change | 0.38 (16.180) | -8.92 (16.945)

26. Other Pre Specified Outcome: Percent Change From Baseline to Week 24 in apoB
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for apoB. Baseline was defined as the last value prior to first dose of study drug. Percent change from baseline was calculated as: [(apoB value at Week 24 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Observed data was used for the analysis, no imputation for the missing data was performed
Time Frame: Baseline; Week 24
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 699 | 1381
percent change | 4.8 (20.41) | -7.1 (20.01)

27. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in apoB
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for apoB. Baseline was defined as the last value prior to first dose of study drug. Percent change from baseline was calculated as: [(apoB value at Week 52 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Observed data was used for the analysis, no imputation for the missing data was performed.
Time Frame: Baseline; Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 676 | 1342
percent change | 3.4 (20.24) | -6.0 (22.54)

28. Other Pre Specified Outcome: Percent Change From Baseline to Week 24 in hsCRP
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for hsCRP. Baseline was defined as the last value prior to first dose of study drug. Percent change from baseline was calculated as: [(hsCRP value at Week 24 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Observed data was used for the analysis, no imputation for the missing data was performed.
Time Frame: Baseline; Week 24
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 706 | 1392
percent change | 2.727 [-33.028 to 59.016] | -16.382 [-51.329 to 34.436]

29. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in hsCRP
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for hsCRP. Baseline was defined as the last value prior to first dose of study drug. Percent change from baseline was calculated as: [(hsCRP value at Week 52 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Observed data was used for the analysis, no imputation for the missing data was performed.
Time Frame: Baseline; Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 681 | 1358
percent change | 1.818 [-36.508 to 60.952] | -14.445 [-50.000 to 43.889]

30. Other Pre Specified Outcome: Percentage of Participants Achieving LDL-C <70 mg/dL at Week 12, 24, and 52
Description: The percentage of participants who achieved lowering in lipid values of LDL-C below 70 mg/dL have been reported. Baseline was defined as the mean of the values at screening (Week -2) and predose Day 1/Week 0. Observed data was used for the analysis, no imputation for the missing data was performed.
Time Frame: Week 12, Week 24, and Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 742 | 1488
Percentage of participants
  Week 12: number analyzed (Participants) | 725 | 1424
  Week 12 | 9.0 | 32.4
  Week 24: number analyzed (Participants) | 707 | 1397
  Week 24 | 10.2 | 32.0
  Week 52: number analyzed (Participants) | 685 | 1364
  Week 52 | 9.5 | 28.2
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to approximately 52 weeks
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began or worsened in severity after the first dose of double-blind study drug and up to 30 days after receiving the last dose of double-blind study drug, were collected and reported.
Arm/Group | Bempedoic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 13/1487 | 2/742
Serious Adverse Events (participants affected / at risk) | 216/1487 | 104/742
Other Adverse Events (participants affected / at risk) | 792/1487 | 381/742
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bempedoic Acid (N=1487) | Placebo (N=742)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 11 | 5
Angina pectoris (Cardiac disorders) | 11 | 6
Angina unstable (Cardiac disorders) | 18 | 12
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 7 | 1
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 2
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 5 | 3
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 4 | 1
Coronary artery disease (Cardiac disorders) | 9 | 6
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dilatation (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 4 | 1
Myocardial infarction (Cardiac disorders) | 8 | 5
Pericarditis (Cardiac disorders) | 2 | 0
Sinus node dysfunction (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Ventricular fibrillation (Cardiac disorders) | 2 | 1
Myotonic dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 1
Goitre (Endocrine disorders) | 1 | 0
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Internal hernia (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis relapsing (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 0 | 1
Eye complication associated with device (General disorders) | 0 | 1
Granuloma (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pelvic mass (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 7 | 4
Vascular stent restenosis (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Immune system disorder (Immune system disorders) | 1 | 0
Abscess jaw (Infections and infestations) | 0 | 1
Abdominal sepsis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 3 | 0
Diverticulitis (Infections and infestations) | 4 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1
Implant site infection (Infections and infestations) | 0 | 1
Infected bite (Infections and infestations) | 1 | 0
Infective aneurysm (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Localised infection (Infections and infestations) | 1 | 0
Medical device site joint infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Salmonella bacteraemia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal osteomyelitis (Infections and infestations) | 1 | 0
Tonsillitis bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 2 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Carotid artery disease (Nervous system disorders) | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 2
Cerebral infarction (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 3
Transient ischaemic attack (Nervous system disorders) | 3 | 2
Major depression (Psychiatric disorders) | 0 | 1
Intensive care unit delirium (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 2 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aortic aneurysm (Vascular disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 2 | 1
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 3
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Enteritis necroticans (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bempedoic Acid (N=1487) | Placebo (N=742)
Anaemia (Blood and lymphatic system disorders) | 41 | 15
Angina pectoris (Cardiac disorders) | 24 | 19
Nausea (Gastrointestinal disorders) | 43 | 19
Constipation (Gastrointestinal disorders) | 26 | 18
Diarrhoea (Gastrointestinal disorders) | 60 | 30
Bronchitis (Infections and infestations) | 52 | 19
Lower respiratory tract infection (Infections and infestations) | 41 | 19
Fatigue (General disorders) | 38 | 25
Sinusitis (Infections and infestations) | 26 | 18
Nasopharyngitis (Infections and infestations) | 146 | 87
Urinary tract infection (Infections and infestations) | 70 | 47
Upper respiratory tract infection (Infections and infestations) | 72 | 31
Blood creatine phosphokinase increased (Investigations) | 35 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 32 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 64 | 44
Back pain (Musculoskeletal and connective tissue disorders) | 55 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 62 | 20
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 30 | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 89 | 45
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 40 | 19
Dizziness (Nervous system disorders) | 65 | 31
Pain in extremity (Musculoskeletal and connective tissue disorders) | 50 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 23
Headache (Nervous system disorders) | 45 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 16
Hypertension (Vascular disorders) | 42 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that that publication be withheld.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT02666664/SAP_000.pdf
  • Study Protocol (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT02666664/Prot_001.pdf